CLINICAL TRIAL: NCT02324049
Title: A Phase I/II Open Label Study in MPS IIIB Subjects to Investigate the Safety, Pharmacokinetics, and Pharmacodynamics/Efficacy of SBC-103 Administered Intravenously
Brief Title: Safety, Pharmacokinetics, and Pharmacodynamics/Efficacy of SBC-103 in Mucopolysaccharidosis III, Type B (MPS IIIB)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NGLU-CL02
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Results first posted 2018-07-12 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Mucopolysaccharidosis IIIB
Keywords: MPS IIIB; Mucopolysaccharidosis; Mucopolysaccharidosis type IIIB; Sanfilippo Syndrome; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn; Carbohydrate Metabolism, Inborn Errors; Connective Tissue Diseases; Lysosomal Storage Diseases; Mucinoses; Mucopolysaccharidoses; Pathologic Processes
MeSH Terms: conditions — Mucopolysaccharidosis III; Mucopolysaccharidoses; Metabolism, Inborn Errors; Metabolic Diseases; Genetic Diseases, Inborn; Carbohydrate Metabolism, Inborn Errors; Connective Tissue Diseases; Lysosomal Storage Diseases; Mucinoses; Pathologic Processes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SBC-103 (Experimental): Part A (Initial therapy): Participants received SBC-103, 0.3, 1.0, or 3.0 mg/kg QOW for 24 weeks, followed by a ≥ 4-week treatment break. Participants enrolled in the lowest dosage first.
  Part B: Participants were escalated to the next highest dose that was considered safe (1.0 or 3.0 mg/kg QOW) for ≥ 8 weeks. Participants who received doses of 0.3 mg/kg in Part A were considered for a second dose escalation to 3.0 mg/kg at any time during Part B provided that they tolerated at least 2 doses of 1.0 mg/kg in Part B. Participants who received and tolerated at least 4 doses of SBC-103 QOW at 3.0 mg/kg were considered for participation in Part C.
  Part C: Participants received SBC-103 5.0 or 10.0 mg/kg administered IV QOW. Dosing in Part C began at the 5.0 mg/kg dose level. The decision to begin dosing the first participant at 10.0 mg/kg was based on the review of safety data at 5.0 mg/kg.
  Interventions: Drug: SBC-103

INTERVENTIONS:
Drug: SBC-103
  Other Names: recombinant human alpha-N-acetylglucosaminidase

SUMMARY:
Study to evaluate the safety and tolerability of intravenous (IV) administration of SBC-103 in participants with mucopolysaccharidosis III, type B (MPS IIIB, Sanfilippo B) with evaluable signs or symptoms of developmental delay.

DETAILED DESCRIPTION:
This study was designed as a 3-part study to evaluate the safety and tolerability of IV administration of SBC-103. Participants enrolled in Part A (0.3, 1.0, or 3.0 milligrams [mg] per kilogram [kg] of SBC-103 administered every other week [QOW] for 24 consecutive weeks). Participants who completed Part A were eligible for Part B (an increase to 1.0 or 3.0 mg/kg QOW). Participants who completed Part B were eligible for Part C (5.0 and/or 10.0 mg/kg to continue through Week156; no participants received both 5.0 and 10.0 mg/kg). Due to the early termination of the SBC-103 development program, including this study, all participants withdrew from Part C at the sponsor's decision. As a result of the early termination of this program, this report provides only safety data.

ELIGIBILITY:
Key Inclusion Criteria:

* A participant was greater than or equal to 2 years of age but less than 12 years of age at the time of informed consent.
* Definitive diagnosis of MPS IIIB.
* Documented developmental delay.

Key Exclusion Criteria:

* Received treatment with gene therapy at any time.
* Previous hematopoietic stem cell or bone marrow transplant.
* Had any internal or non-removable external metal items that presented a safety risk for study assessments that utilized magnetic fields, or any other medical condition or circumstance in which magnetic resonance imaging was contraindicated according to local institutional policy.
* Known hypersensitivity to eggs.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (2):
  - Minneapolis, Minnesota
  - Pittsburgh, Pennsylvania
- Barcelona, Spain
- Birmingham, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Diagnosis of mucopolysaccharidosis III, type B (MPS IIIB), determined by either documented deficiency in Alpha-N-acetylglucosaminidase (NAGLU) enzyme activity ≤10% of the mean value in normal individuals at Screening OR documented functionally-relevant mutations in both alleles of the NAGLU gene based on historical or Screening laboratory results.
Groups:
- SBC-103: Part A (Initial therapy): Participants received SBC-103, 0.3, 1.0, or 3.0 milligrams (mg) per kilogram (kg) every other week (QOW) for 24 weeks, followed by a ≥ 4-week treatment break. Participants enrolled in the lowest dosage first.
  Part B: Participants were escalated to the next highest dose that was considered safe (1.0 or 3.0 mg/kg QOW) for ≥ 8 weeks. Participants who received doses of 0.3 mg/kg in Part A were considered for a second dose escalation to 3.0 mg/kg at any time during Part B provided that they tolerated at least 2 doses of 1.0 mg/kg in Part B. Participants who received and tolerated at least 4 doses of SBC-103 QOW at 3.0 mg/kg were considered for participation in Part C.
  Part C: Participants received SBC-103 5.0 or 10.0 mg/kg administered intravenous (IV) QOW. Dosing in Part C began at the 5.0 mg/kg dose level. The decision to begin dosing the first participant at 10.0 mg/kg was based on the review of safety data at 5.0 mg/kg.
Period: Part A
Arm/Group | SBC-103
Started | 11
Safety Analysis Set | 11 (Participants with informed consent, confirmed MPS IIIB diagnosis, and received any amount of SBC-103)
Completed | 11
Not Completed | 0
Period: Part B
Arm/Group | SBC-103
Started | 11
Safety Analysis Set | 11
Completed | 11
Not Completed | 0
Period: Part C
Arm/Group | SBC-103
Started | 11
Safety Analysis Set | 11
Completed | 0
Not Completed | 11
Not completed — Study terminated | 11

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants for whom informed consent had been obtained, who had a confirmed diagnosis of MPS IIIB, and who had received any amount of SBC-103.
Arm/Group | SBC-103
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1
Overall Age at Diagnosis [Median (Full Range); unit: Months] — Population: There were 5 participants in the 5.0 mg/kg group and 6 participants in the 10.0 mg/kg group.
  Months
    5.0 mg/kg: number analyzed (Participants) | 5
    5.0 mg/kg | 48.0 [18 to 57]
    10.0 mg/kg: number analyzed (Participants) | 6
    10.0 mg/kg | 25.0 [12 to 77]
    Overall | 37.0 [12 to 77]

OUTCOME MEASURES:

1. Primary Outcome: Number Of Participants Who Experienced Severe Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event (AE) that occurred after administration of the first dose of study drug on Day 1 (Part A). A severe AE was defined as an AE that was incapacitating and required medical intervention. TEAEs were summarized cumulatively over the entire study and separately for Part C, data for all severe TEAEs throughout the entire study is presented. A summary of serious and all other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline to Week 142
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SBC-103
Number analyzed (Participants) | 11
Participants
  5.0 mg/kg | 1
  10.0 mg/kg | 0
  Overall | 1

ADVERSE EVENTS:
Time Frame: Day 1 postdose up to Week 142
Arm/Group | SBC-103
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBC-103 (N=11)
Bacteraemia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Cyanosis (Cardiac disorders) | 1
Pyrexia (General disorders) | 1
Blood pressure increased (Investigations) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SBC-103 (N=11)
Pyrexia (General disorders) | 9
Catheter site erythema (General disorders) | 2
Catheter site rash (General disorders) | 1
Catheter site swelling (General disorders) | 1
Influenza like illness (General disorders) | 1
Local swelling (General disorders) | 1
Pain (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 4
Lower respiratory tract infection (Infections and infestations) | 2
Rhinitis (Infections and infestations) | 2
Gastroenteritis viral (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Pharyngitis streptococcal (Infections and infestations) | 1
Candida nappy rash (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Eye infection bacterial (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oral herpes (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Paronychia (Infections and infestations) | 1
Respiratory tract infection viral (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 4
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin plaque (Skin and subcutaneous tissue disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 6
Salivary hypersecretion (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Breath odour (Gastrointestinal disorders) | 1
Eructation (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Pancreatic enlargement (Gastrointestinal disorders) | 1
Swollen tongue (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Head injury (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Anaesthetic complication neurological (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Eye contusion (Injury, poisoning and procedural complications) | 1
Eyelid injury (Injury, poisoning and procedural complications) | 1
Foreign body (Injury, poisoning and procedural complications) | 1
Lip injury (Injury, poisoning and procedural complications) | 1
Mouth injury (Injury, poisoning and procedural complications) | 1
Cardiac murmur (Investigations) | 2
Body temperature increased (Investigations) | 1
CSF protein increased (Investigations) | 1
Electrocardiogram Q wave abnormal (Investigations) | 1
Liver palpable (Investigations) | 1
Mean platelet volume increased (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Serum ferritin decreased (Investigations) | 1
Deafness (Ear and labyrinth disorders) | 4
Ear pain (Ear and labyrinth disorders) | 2
Deafness bilateral (Ear and labyrinth disorders) | 1
Hypoacusis (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Flushing (Vascular disorders) | 2
Hyperaemia (Vascular disorders) | 2
Hypertension (Vascular disorders) | 2
Headache (Nervous system disorders) | 1
Hyperreflexia (Nervous system disorders) | 1
Hypertonia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 1
Psychomotor hyperactivity (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Left ventricular hypertrophy (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Mydriasis (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Muscle mass (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Iron deficiency (Metabolism and nutrition disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Dysmorphism (Congenital, familial and genetic disorders) | 1
Precocious puberty (Endocrine disorders) | 1
Device occlusion (Product Issues) | 1
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Hypervigilance (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 2
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/49/NCT02324049/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT02324049/SAP_001.pdf